CLINICAL TRIAL: NCT02523781
Title: Evaluation of an Information Pamphlet to Improve Knowledge Concerning the Impacts and the Importance of Healthy Lifestyle After a Pregnancy With Hypertension
Brief Title: Evaluation of an Information Pamphlet for Postpartum Women That Had a Hypertensive Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nadine Sauvé, Researcher of the Mother-Child axis of the CRCHUS, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1099
Record Dates: First submitted 2015-07-30; First posted 2015-08-14 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: preeclampsia; information pamphlet; patient education
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group does not receive the information pamphlet
- Intervention group (Experimental): The intervention group receives the information pamphlet
  Interventions: Other: information pamphlet

INTERVENTIONS:
Other: information pamphlet — The intervention group receives the information pamphlet
  Arms: Intervention group

SUMMARY:
It is known that preeclampsia is a risk factor for cardiovascular diseases, diabetes, chronic hypertension, nephropathy and thromboembolism. The study's aim, subsequent to these informations, is to help prevent those consequences. Information tools have been known to enhance retention of information given orally. The objective of this study is to assess the knowledge and satisfaction of women after an episode of preeclampsia after reading an explanatory pamphlet on preeclampsia. The investigators also want to change their perception on cardiovascular risk, their risk of recurrence and preeclampsia's medium to long-term consequences and the ways to prevent them.

DETAILED DESCRIPTION:
This is a randomised-controlled trial. Women recruted will first answer a questionnaire assessing demographic data, knowledge about risks in the future, perception of cardiovascular risk, anxiety about that risk and satisfaction about information received or collected.

Then, women in the intervention group will receive the pamphlet. One month after, women in both groups will receive a questionnaire similar to the first one assessing knowledge about risks in the future, perception of cardiovascular risk, anxiety about that risk and satisfaction about information received or collected, including the pamphlet for the intervention group.

The pamphlet was validated by a multidisciplany team including patients, doctors, nurses, education specialists and communication specialists.

The questionnaire was also validated by the same multidisciplinary team. Section on knowledge and anxiety were remodeled from previously validated questionnaires Section on perception of cardiovascular risk was reproduced and translated with permission from its author.

Section on satisfaction was reproduced from the investigators' previous study where it was validated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* followed at the CHUS obstetrical clinic for a 4 weeks to 18 months postpartum follow up
* had hypertension in her last pregnancy

Exclusion criteria:

* Not able to read and write in French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
knowledge improvement (questionnaire with check list and true/false questions). | 4 weeks
  The primary outcome will be the comparison of knowledge between the intervention (with the pamphlet) and the control (without the pamphlet) group at one month with a validated questionnaire (knowledge: check list and true/false questions).

SECONDARY OUTCOMES:
Perception of cardiovascular risk between the intervention and the control group at one month (Likert scale) | 4 weeks
  The comparison of perception of cardiovascular risk at one month between the intervention (with the pamphlet) and the control (without the pamphlet) group with a validated Likert scale included in the questionnaire.
Anxiety between the intervention and the control group at one month.(Likert scale) | 4 weeks
  Comparison of anxiety at one month between the intervention and the control group with a validated Likert scale included in the questionnaire.
Satisfaction between the intervention and the control group at one month.(Likert scale) | 4 weeks
  Comparison of satisfaction about all sources of information at one month between the intervention and the control group with a validated Likert scale included in the questionnaire.
Perception of cardiovascular risk in the intervention group between baseline and at one month (Likert scale) | 4 weeks
  The comparison of perception of cardiovascular risk between baseline and at one month in the intervention group with a validated Likert scale included in the questionnaire.
Perception of cardiovascular risk between baseline and at one month in the control group. (Likert scale) | 4 weeks
  The comparison of perception of cardiovascular risk between baseline and at one month in the control group with a validated Likert scale included in the questionnaire.
Anxiety in the intervention group between baseline and at one month (Likert scale) | 4 weeks
  The comparison of anxiety between baseline and at one month in the intervention group with a validated Likert scale included in the questionnaire.
Anxiety in the control group between baseline and at one month (Likert scale) | 4 weeks
  The comparison of anxiety between baseline and at one month in the control group with a validated Likert scale included in the questionnaire
Satisfaction in the intervention group between baseline and at one month(Likert scale) | 4 weeks
  The comparison of satisfaction between baseline and at one month in the intervention group with a validated Likert scale included in the questionnaire.
Satisfaction in the control group between baseline and at one month (Likert scale) | 4 weeks
  The comparison of satisfaction between baseline and at one month in the control group with a validated Likert scale included in the questionnaire.
Knowledge in the intervention group between baseline and at one month (questionnaire with check list and true/false questions). | 4 weeks
  The comparison of baseline knowledge and knowledge at one month in the intervention group with a validated questionnaire (knowledge: check list and true/false questions).
Knowledge in the control group between baseline and at one month (questionnaire with check list and true/false questions). | 4 weeks
  The comparison of Baseline knowledge and knowledge at one month in the control group with a validated questionnaire (knowledge: check list and true/false questions).

CONTACTS AND LOCATIONS:
Overall Officials: Sauvé Nadine, MD, Principal Investigator — Université de Sherbrooke; Anne-Marie côté, MD, Study Chair — Université de Sherbrooke; Annabelle Cumyn, MD, Study Chair — Université de Sherbrooke; Marie-Eve Roy-Lacroix, MD, Study Chair — Université de Sherbrooke; Myriam Champagne, MD, Study Chair — Université de Sherbrooke; Marie-Hélène Pesant, MD, Study Chair — Université de Sherbrooke
Locations (1):
- Centre Hopitalier Universiatire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No